CLINICAL TRIAL: NCT03528317
Title: Alternate Day Fasting Combined With a High Protein Background Diet for Weight Loss and Weight Maintenance in Adults With Obesity
Brief Title: Alternate Day Fasting Combined With a High Protein Background Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Krista Varady, Professor of Nutrition, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1363
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alternate day fasting (Experimental): Alternate day fasting with a high protein diet
  Interventions: Other: Alternate day fasting

INTERVENTIONS:
Other: Alternate day fasting — Alternate day fasting with a high protein diet

SUMMARY:
The aims of this study are as follows: AIM 1: To examine the weight loss and weight maintenance efficacy of an alternate day fasting-high protein (ADF-HP) diet; AIM 2: To examine the effects of an ADF-HP diet on metabolic disease risk factors (plasma lipids, fasting glucose, fasting insulin, insulin resistance).

DETAILED DESCRIPTION:
Background: Accumulating evidence suggests that alternate day fasting (ADF) is an effective diet strategy to help individuals with obesity lose weight and lower metabolic disease risk. ADF regimens include a "feast day" where food is consumed ad-libitum over 24 h, alternated with a "fast day" where intake is limited to ~600 kcal over 24 h. What has yet to be elucidated is whether consuming a high protein diet (as meal replacements) during ADF is effective for weight loss, weight maintenance, and metabolic disease risk reduction in individuals with obesity.

Objective: The aims of this study are as follows: AIM 1: To examine the weight loss and weight maintenance efficacy of an alternate day fasting-high protein (ADF-HP) diet; AIM 2: To examine the effects of an ADF-HP diet on metabolic disease risk factors (plasma lipids, fasting glucose, fasting insulin, insulin resistance).

Methods: A 24-week, single-center, longitudinal pilot study will be conducted to test the study objectives. The trial will be divided into 2 consecutive intervention periods: (1) 12-week weight loss period, and (2) 12-week weight maintenance period. Subjects with obesity will participate in an ADF-HP: alternate day fasting-high protein diet: 600 kcal "fast day" alternated with ad libitum "feast day", 35% kcal as protein. ADF-HP subjects will consume the Optifast HP Shake Mix (Nestle) on each day of the trial. Body weight, insulin, glucose, and insulin resistance, will be measured at baseline, week 12, and week 24.

Significance: These findings may show that alternate day fasting combined with high protein meal replacements may be implemented as an effective diet therapy to help individuals with obesity lose weight, maintain weight loss, and sustain reductions in metabolic disease risk.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65 years old
* BMI between 30.0 and 49.9 kg/m2
* Previously sedentary or lightly active

Exclusion Criteria:

* Diabetic
* History of binge eating disorder
* Taking weight loss-inducing medications
* Not weight stable for 3 months prior to the study (weight gain or loss > 4 kg)
* Perimenopausal or have an irregular menstrual cycle (menses that does not appear every 27-32 days)
* Pregnant or trying to become pregnant
* Night shift worker
* Smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Body weight | Change from baseline to week 24
  Measured by digital scale

SECONDARY OUTCOMES:
Triglycerides | Change from baseline to week 24
  Measured by ELISA
Glucose | Change from baseline to week 24
  Measured by glucometer
Insulin | Change from baseline to week 24
  Measured ELISA
Insulin resistance | Change from baseline to week 24
  Measured as HOMA-IR
Sleep quality | Change from baseline to week 24
  Measured by Pittsburgh Sleep Quality Index (PSQI), total score of 0-21. A PSQI
Insomnia severity | Change from baseline to week 24
  Measured by Insomnia Severity Index (ISI), total score of 0-28. The total score for the ISI is interpreted as follows: no clinically significant insomnia (0-7), sub-threshold insomnia (8-14), moderate severity insomnia (15-21), and severe insomnia (22-28).
Sleep apnea | Change from baseline to week 24
  Measured by Berlin Questionnaire, measures the presence or absence of sleep apnea
Appetite | Change from baseline to week 24
  Measured by Visual analog scale (VAS). Scored from 0-100. Higher score means higher appetite.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Varady, Principal Investigator — University of Illinois Chicago (UIC)
Locations (1):
- University of Illinois, Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akasheh RT, Fantuzzi G, Varady KA, Cheng TD, Kalam F. Reduced Serum PD-L1 and Markers of Inflammation in Response to Alternate Day Fasting With a Low-Carbohydrate Intervention: A Secondary Analysis of a Single-Arm Trial. Curr Dev Nutr. 2025 Feb 14;9(3):104566. doi: 10.1016/j.cdnut.2025.104566. eCollection 2025 Mar. PMID 40145019
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Kalam F, Gabel K, Cienfuegos S, Wiseman E, Ezpeleta M, Pavlou V, Varady KA. Changes in subjective measures of appetite during 6 months of alternate day fasting with a low carbohydrate diet. Clin Nutr ESPEN. 2021 Feb;41:417-422. doi: 10.1016/j.clnesp.2020.10.007. Epub 2020 Oct 29. PMID 33487299
- [Derived] Lin S, Lima Oliveira M, Gabel K, Kalam F, Cienfuegos S, Ezpeleta M, Bhutani S, Varady KA. Does the weight loss efficacy of alternate day fasting differ according to sex and menopausal status? Nutr Metab Cardiovasc Dis. 2021 Feb 8;31(2):641-649. doi: 10.1016/j.numecd.2020.10.018. Epub 2020 Oct 31. PMID 33358713